CLINICAL TRIAL: NCT05402241
Title: Isolated Restricted Diffusion at Admission Predicts Survival in Patients of Glioblastoma Multiforme (IRD GBM)- A Prospective Pilot Study
Brief Title: IRD at Admission Predicts Survival of GBM Patients - a Prospective Pilot Study
Acronym: IRD-GBM
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Collaborators: CancerCare Manitoba (Other)
Responsible Party: Sponsor
Other Study IDs: 1
Record Dates: First submitted 2021-10-22; First posted 2022-06-02 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-01

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma, Multiforme; Isolated Restricted Diffusion foci
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Glioblastomas (GBM) are the most common primary malignant brain tumor with a very high recurrence rate and an average survival of 14 months. Identifying an imaging biomarker to predict recurrence is critical. Using a special MRI technique called diffusion weighted imaging (DWI), a recent retrospective study described isolated restricted diffusion (IRD) foci. The presence of IRD was found in 40% of patients with GBM on index imaging and was associated with longer survival. IRD foci are not currently identified as having a tumor focus and are not included in treatment strategies and guidelines. These findings need to be confirmed in a prospective study. The investigators propose a prospective pilot study to establish the incidence of IRD on the index imaging of patients with GBM. The investigators will collect surgical samples from these foci to establish the histological and molecular signature to confirm GBM in these newly identified foci. The results from this pilot study will guide the planning of a larger well powered multicenter study that will help establish IRD as an imaging biomarker in the GBM management guidelines, which will help improve the outcomes in patients with GBM.

DETAILED DESCRIPTION:
Glioblastomas (GBM) are the most common type of primary malignant brain tumor with a very high rate of recurrence. The average survival of patients with GBM is 14 months, and the 5-year survival rate is approximately 4 to 5%. Identifying an imaging biomarker to predict recurrence is critical. Using a special MRI technique called diffusion weighted imaging (DWI), the investigators recently described a focus of isolated restricted diffusion (IRD) in a retrospective study. Presence of IRD was found in 40% of patients with GBM on index imaging and was associated with longer survival. The foci of IRD are not currently identified as having a tumor focus and are not included in treatment strategies and guidelines. The results from this pilot study will help plan for a larger well powered multicenter study that will help establish IRD as an imaging biomarker in the GBM management guidelines. The investigators hypothesize that IRD foci when present, are foci of GBM and when untreated, will be the site of recurrence.

This pilot study will use a prospective cohort study design, to establish the incidence of IRD on the index imaging of participants with GBM. Surgical samples will be collected from these foci to establish the histological and molecular signature to confirm GBM in these newly identified foci. The study population will include patients that present with newly diagnosed with GBM. All newly diagnosed GBM participants will be screened for the study using the study inclusion and exclusion criteria. After the standard of care MRI/DWI is done and reviewed, eligible participants will be approached by the research team, for discussion of the study and potential consent for participation. All participants will undergo further treatment and management as per institutional standard including the clinical and imaging follow up. Each MRI will be screened by experienced neuro-radiologists to identify the presence of isolated restricted diffusion foci. In those participants with isolated restricted diffusion foci on MRI, the neurosurgeon (on for the day) will assess the feasibility and safety of targeted biopsy from this focus. The targeted biopsy will only be considered when it is deemed safe and feasible based on the location and surgical approach, which will be determined by the neurosurgeon. This will reduce any undue risk for research purposes. The biopsy samples will undergo standard of care laboratory histopathological and molecular testing to establish the pathological and molecular signatures of these tumors. The neuropathologic examination will be performed by neuropathologists. Informed consent will be obtained from the patients to participate in the study.

The aim of this study is to establish a new imaging biomarker and to determine its association with known molecular alterations in GBM. The investigators will also explore the incidence of isolated restricted diffusion in GBM participants, the number of IRD foci that proceed to contrast enhancement on follow up, the true number of IRD foci, and the survival pattern of the study participants with isolated restricted diffusion.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Patients with suspected GBM on initial MRI of brain
* MRI scans with isolated restricted diffusion foci noted

Exclusion Criteria:

* Participants who are pregnant
* Known contraindication to MRI contrast agent, e.g., allergy or anaphylactic reaction
* Known end-stage renal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: newly diagnosed patients with GBM
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Incidence of isolated restricted diffusion (IRD) in GBM patients | Upon completion of the study, which will be approximately 2 years
  proportion of GBM participants with IRD
Incidence of IRD foci proceeding to contrast enhancement on 3 month follow up | through completion of the study approximately 2 years
  proportion of participants that have contrast enhancement on 3 month follow-up
Incidence of IRD foci proceeding to contrast enhancement on 6 month follow up | through completion of the study approximately 2 years
  proportion of participants that have contrast enhancement on 6 month on follow-up
Incidence of IRD foci that are from the GMB foci | through completion of the study, approximately 2 years
  proportion of IRD foci that originate from the GBM foci
relationship of molecular alteration with GBM foci and the IRD | Upon completion of the study approximately 2 years
  descriptive analysis
Survival patterns of GBM participants with IRD | Upon completion of the study approximately 2 years
  mortality

CONTACTS AND LOCATIONS:
Overall Officials: Jai Shankar, MD, Principal Investigator — University of Manitoba
Locations (2):
- Canada (2):
  - University of Manitoba, Winnipeg, Manitoba
  - Health Sciences Centre, Winnipeg MB, Manitoba